CLINICAL TRIAL: NCT05575869
Title: Evaluate the Impact of Online Educational Material (PRONEtect Educational Hub) on Nursing Students' Knowledge, Confidence Levels, and Application of Knowledge Regarding Skin Protection of the Prone Ventilated Patient - a Randomised Controlled Study
Brief Title: Evaluation of the Impact of the PRONEtect Education Hub vs. Classic Lecture, on the Competencies of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PRONEtection #2
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Prone Position; Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The lecturers at the nursing schools (x2) will have no access to the results of the surveys. A study number is assigned to the students and with the study number they enter their answers to the questionnaires
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Access to online PRONEtect educational material (Experimental): A website with educational material (simulation video, protocol, checklist).
  Interventions: Other: (online) PRONEtect educational material
- Control group: Classic one-hour lecture (Active Comparator): Didactive presentation by the usual nursing school lecturer.
  Interventions: Other: Classic (normal) one hour lesson/lecture

INTERVENTIONS:
Other: (online) PRONEtect educational material — This is a website containing educational material like short simulation videos on how to turn a patient from supine-to-prone and prone-to-supine positioning, how to protect the skin from incontinence, or before securing endotracheal-/nasogastric tubes, how to reposition the patient to prevent pressure injuries, a full protocol regarding prone positioning etc.
  Arms: Experimental group: Access to online PRONEtect educational material
Other: Classic (normal) one hour lesson/lecture — As per normal, a classroom lecture given by the nursing school by one of the nursing school lecturers.
  Arms: Control group: Classic one-hour lecture

SUMMARY:
The goal of this randomised controlled trial is to compare the impact of online educational material versus a classic lecture on the confidence levels, knowledge and knowledge application of final-year nursing students.

Participants will be asked to complete a baseline self-efficacy evaluation and a baseline knowledge test which were validated by the 11-member international expert panel previously established.

After randomization, the control group will be asked to attend a classic 1-hour lecture at the nursing school about the topic of prone positioning and skin/tissue damage prevention.

The experimental group will get access to the PRONEtect educational website containing short simulation videos and other learning materials.

Three weeks later the participants will be asked to complete the self-efficacy evaluation and knowledge assessment again, additionally a knowledge application assessment.

All the questionnaires will be administered via Qualtrics.

ELIGIBILITY:
Inclusion Criteria:

* Final year nursing students studying towards their Bachelor in Nursing degree
* Chosen topics of critical care nursing as supplementary subject or critical care subjects as part of their course or complex wound management as part of their course.

Exclusion Criteria:

Nursing students who are not yet in their final year of studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Knowledge assessment (test score) | 3 weeks
  A total sample size of 78 participants (39 in each group, 1:1 allocation ratio) to have at least 80% power to demonstrate non-inferiority of the online package (experimental group) compared to the classical lecture (control group) with respect to the mean change from baseline in knowledge at week 3 at the one-sided 1.25% significance level, when the non-inferiority margin is set at 1 point and when we assume a common standard deviation in both groups of 2.5 points, a true difference between the groups of 1 point in favor of the online package, and a drop-out rate of 20%.

SECONDARY OUTCOMES:
Confidence levels (survey scores) | 3 weeks
  A total sample size of 78 participants (39 in each group, 1:1 allocation ratio) to have at least 80% power to demonstrate non-inferiority of the online package (experimental group) compared to the classical lecture (control group) with respect to the mean change from baseline in knowledge at week 3 at the one-sided 1.25% significance level, when the non-inferiority margin is set at 1 point and when we assume a common standard deviation in both groups of 2.5 points, a true difference between the groups of 1 point in favor of the online package, and a drop-out rate of 20%.
Difference between the "Knowledge application" (test score) between the groups | 3 weeks
  Difference between the "Knowledge application" (test score) of 1-2 points between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fourie A, Ahtiala M, Black J, Campos HH, Coyer F, Gefen A, LeBlanc K, Smet S, Vollman K, Walsh Y, Karlberg-Traav M, Beeckman D. Enhancing prone positioning and skin damage prevention education: A randomized controlled non-inferiority trial comparing a digital education hub (PRONEtect) and a traditional lecture on final-year nursing participants' confidence and knowledge. J Tissue Viability. 2024 May;33(2):298-304. doi: 10.1016/j.jtv.2024.02.008. Epub 2024 Feb 19. PMID 38402096